CLINICAL TRIAL: NCT07061522
Title: Investigation of the Impact of Smoking Addiction on the Speed and Coordination of Lower Extremity Movements
Brief Title: Effects of Smoking Addiction on Lower Limb Speed and Coordination
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: Smoking Add-Coordination-1
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking Addiction Group: Participants in this group will be individuals who meet the criteria for smoking addiction based on both the DSM-IV-TR criteria and the Fagerström Test for Nicotine Dependence. They must have smoked at least one cigarette per day for the past 12 months.
  Interventions: Other: Behavioral/Physical Assessment
- Non-Smokers: Participants in this group will be healthy individuals aged 18-25 with no history of smoking within the past year. They will be matched in terms of age and BMI to the smoking group and will serve as the control cohort.
  Interventions: Other: Behavioral/Physical Assessment

INTERVENTIONS:
Other: Behavioral/Physical Assessment — This study will not include any therapeutic or clinical intervention. Instead, participants will undergo a series of structured physical and questionnaire-based assessments to evaluate lower extremity motor performance. These include the Fagerström Test for Nicotine Dependence and DSM-IV-TR criteria to classify smoking addiction. Anthropometric measurements such as Body Mass Index (BMI) and bimalleolar diameter/circumference will be recorded to assess potential confounding structural factors. Lower extremity coordination will be evaluated using the Lower Extremity Motor Coordination Test (LEMOCOT), and movement speed will be assessed with a 30-meter sprint test. All assessments will be conducted once in a controlled laboratory setting and are intended solely for comparative analysis between smokers and non-smokers.

SUMMARY:
This observational case-control study will investigate the impact of smoking addiction on lower extremity speed and coordination in young adults. Participants aged 18-25 will be divided into two groups based on their smoking status. The study will compare motor coordination and sprint performance between smokers and non-smokers using objective physical tests under standardized laboratory conditions.

DETAILED DESCRIPTION:
This non-randomized controlled study will aim to evaluate the effects of smoking addiction on the speed and coordination of lower extremity movements among healthy young adults. Smoking is known to have detrimental effects on vascular, musculoskeletal, and neurological systems, yet its impact on motor performance-particularly in the lower limbs-has not been sufficiently studied.

Participants aged 18-25 will be categorized into smoker and non-smoker groups based on DSM-IV-TR nicotine dependence criteria and the Fagerström Test. The Lower Extremity Motor Coordination Test (LEMOCOT) will be used to assess motor coordination, while a 30-meter sprint test will evaluate movement speed. Additionally, body mass index (BMI) and bimalleolar diameter and circumference will be recorded to control for confounding physical variables.

All assessments will be conducted in a controlled laboratory environment. The results will be analyzed to determine whether smoking addiction is associated with impaired lower limb motor function. The findings may provide new insights into the functional consequences of smoking in young adults and contribute to the design of preventive and rehabilitative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Smoking ≥1 cigarette daily for at least 12 months
* Age between 18-25
* Literate and cooperative
* BMI: 18.5-29.9 kg/m²

Exclusion Criteria:

* Orthopedic, neurological, or neuromuscular conditions impairing walking
* Chronic pulmonary or cardiac disease
* Cognitive impairment
* BMI ≥30 kg/m²

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults aged 18-25 who are either current smokers (according to DSM-IV-TR criteria) or non-smokers. Participants must be physically active enough to perform sprint and coordination tasks, with BMI within a defined range (18.5-29.9 kg/m²). Participants are recruited from a university setting using both institutional announcements and snowball sampling.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Coordination Score | Baseline
  Tool: LEMOCOT (Lower Extremity Motor Coordination Test) Description: Total number of valid taps within 20 seconds.
Sprint Time | Baseline
  Tool: 30-Meter Sprint Test Description: Time in seconds taken to complete a 30-meter run at maximum speed.

SECONDARY OUTCOMES:
Nicotine Dependence Score | Baseline
  Tool: Fagerström Test for Nicotine Dependence Description: Total score assessing severity of nicotine addiction.
BMI (Body Mass Index) | Baseline
  Calculated as weight (kg)/height² (m²), to assess weight-related influence on movement.
Bimalleolar Diameter and Circumference | Baseline
  Measured with caliper and tape to assess potential structural differences affecting motor coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)